CLINICAL TRIAL: NCT01926795
Title: Immobilization Versus Observation in Children With Toddler's Fractures: a Prospective Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prisma Health-Upstate (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00025178
Record Dates: First submitted 2013-08-19; First posted 2013-08-21 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2015-04

CONDITIONS: Tibial Fractures
Keywords: toddler's fracture; tibial fracture; children
MeSH Terms: conditions — Tibial Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Short Leg Cast (Active Comparator): Patient will be placed in a short leg cast for approximately 3 weeks or until radiographic union
  Interventions: Procedure: Short leg cast
- No immobilization (Experimental): No cast or splint will be applied to the injured extremity
  Interventions: Procedure: No Immobilization
- Observational (Other): Patient will be treated based on the parents comfort. This arm will consist of individuals in which the parent/guardian did not agree to randomization, but did consent for observational follow-up regardless of treatment.
  Interventions: Procedure: Short leg cast; Procedure: No Immobilization

INTERVENTIONS:
Procedure: Short leg cast
  Arms: Observational; Short Leg Cast
Procedure: No Immobilization
  Arms: No immobilization; Observational

SUMMARY:
Toddler's fractures of the tibia are by definition non-displaced and of a stable pattern. Children have thickened periosteum compared with adults, which therefore may impart stability to the fracture without the need for additional immobilization. The goal of the study is to evaluate whether or not there is a difference in children treated with and without cast immobilization in regards to time to ambulation; perceived pain; difficulty in dressing & bathing; radiographic displacement or angulation; and time missed from work or daycare. Our null hypothesis is that there will be no difference in clinical or radiographic outcomes between the groups.

ELIGIBILITY:
Inclusion Criteria:

* • Children ages 1-5 years old with radiographic evidence of a non-displaced spiral or oblique fracture of the tibial shaft or metaphysis.

Exclusion Criteria:

* • Children with clinical suspicion but lack of radiographic evidence for toddler's fracture

  * Fractures displaced >2mm
  * Open fractures
  * Pathologic fracture
  * Fractures involving the physis
  * Previous fracture of the ipsilateral extremity
  * Concomitant fracture involving the ipsilateral or contralateral leg
  * Concomitant head injury
  * Non-ambulatory children (i.e., those who have not yet begun to walk)
  * Children with bone-metabolism disorders (i.e., osteogenesis imperfect, rickets)
  * Children who are geographically prohibited from following up in our system
  * Children whose caregivers are not proficient in English
  * Presentation >7 days from injury
  * Cases considered to be non-accidental trauma

Ages: 1 Year to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 21 (Actual)
Dates: Start 2013-06; Primary Completion 2014-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Days to Ambulation | 12 weeks
  Recorded in parent journal, date of first ambulation without assistance.

SECONDARY OUTCOMES:
Fracture displacement | 12 weeks
  Displacement of the fracture greater than 2 mm in any direction.

CONTACTS AND LOCATIONS:
Overall Officials: Michael L Beckish, MD, Principal Investigator — Greenville Hospital System
Locations (1):
- Greenville Hospital System, Greenville, South Carolina, United States